CLINICAL TRIAL: NCT03414021
Title: Quantification in Nuclear Medicine: Interest of the in SPECT-CT Scan SUVspect in Thea New Generation of Gamma-cameras With Semiconductor. Data Collection for the Constitution of an Observatory of Scintigraphies
Brief Title: Interest of the SPECT-CT Scan SUVspect in the New Generation of Gamma-cameras With Semiconductor
Acronym: GAMMA-CAM
Status: Recruiting | Type: Observational
Sponsor: Lille Catholic University (Other)
Responsible Party: Sponsor
Other Study IDs: OBS-0030
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Thyroid Diseases; Heart Diseases; Bone Diseases; Brain Diseases; Kidney Diseases
Keywords: Nuclear Medicine; SPECT-CT Scan; gamma-camera with semiconductor
MeSH Terms: conditions — Thyroid Diseases; Heart Diseases; Bone Diseases; Brain Diseases; Kidney Diseases | interventions — Single Photon Emission Computed Tomography Computed Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Thyroid Diseases: SPECT-CT Scan
  Interventions: Diagnostic Test: SPECT-CT Scan
- Heart Diseases: SPECT-CT Scan
  Interventions: Diagnostic Test: SPECT-CT Scan
- Bone Diseases: SPECT-CT Scan
  Interventions: Diagnostic Test: SPECT-CT Scan
- Brain Diseases: SPECT-CT Scan
  Interventions: Diagnostic Test: SPECT-CT Scan
- Kidney Diseases: SPECT-CT Scan
  Interventions: Diagnostic Test: SPECT-CT Scan

INTERVENTIONS:
Diagnostic Test: SPECT-CT Scan — Injection of a Tracer and SPECT-CT Scan

SUMMARY:
Since 2017, a revolution began in the departments of nuclear medicine, with the routine use of gamma-cameras with semiconductor. These gamma-cameras (which obtained the CE-marking in 2016), offer a technological breakthrough by providing an additional information. They allow "to quantify" for the 1st time in clinical routine conditions, the quantity of radioactivity, by means of a "SUVspect", in a volume of interest, while respecting the recommendations of best practice of the learned societies of French nuclear medicine (SFMN), European (EANM) and American (SNM), without injection of tracer nor acquisition or additional irradiation. The SUVspect is therefore an indicator of the quantity of tracer in a given volume of acquisition.

Until now, the interpretation criteria of scintigraphies are based on the homogeneity of distribution of a tracer in the explored organ (for single organs such as the heart or the thyroid, for example) or in the asymmetry of distribution of the tracer (for the double organs, such as the kidney or the joints).

This new gamma-camera allows to study the distribution of the radio-tracers in "list" mode, allowing to retrospectively reconstruct the images in various ways (for example, by modifying the size of the matrix of acquisition, the energy windows, the time of acquisition). Therefore, we can simulate and propose modifications in current procedures.

Every patient referred to our department of nuclear medicine to undergo a scintigraphy with a tracer of nuclear medicine (with a marketing authorization) can, while benefiting from an examination by this gamma-camera, to be the object of this study, and to profit from this additional information.

So, without changing the diagnosis or the usual care, we wish to take advantage of this additional information to improve the criteria of interpretation of our examinations.

This possibility being new, there is no available bibliography (our department is the 5th department of nuclear medicine in Europe to equip itself with this large field-of-view gamma-camera CZT, the DNM 670, made by General Electric), while 2961 articles speak about the SUVmax (in PET) in Pubmed.

ELIGIBILITY:
Inclusion Criteria:

- informed adult patients referred to our department of nuclear medicine for a nuclear medicine exploration

Exclusion Criteria:

* Refusal to participate
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient referred to our departments of nuclear medicine for a nuclear médicine exploration
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-01-31 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
SUVspect | 5 years
  Pathological threshold (SUVspect) for every type of scintigraphy

SECONDARY OUTCOMES:
Matrix size | 5 years
  Optimize the reconstruction parameters of the images
duration of image acquisition | 5 years
  Optimize the reconstruction parameters of the images

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Blaire, MD, Principal Investigator — GIE HUMANITEP, GHICL; Alban Baillez, MD, Principal Investigator — GIE HUMANITEP, GHICL
Locations (2):
- France (2):
  - Hopital Privé Le Bois, Lille, Hauts-de-France
  - Humanitep, Lomme, Hauts-de-France

IPD SHARING:
Plan to Share IPD: No